CLINICAL TRIAL: NCT03644420
Title: Association Between Preoperative Clinical Evaluation, Radiological Classifications and Histopathology in Patients With Knee Osteoarthritis Receiving a Prosthesis
Brief Title: Evaluation of Patients With Knee Osteoarthritis Receiving a Prosthesis
Acronym: Chondrolike
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Institut de Prévention et de Recherche sur l'Ostéoporose (Unknown)
Responsible Party: Sponsor
Other Study IDs: RT-07
Record Dates: First submitted 2018-07-25; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee; Perfusion; Bone Marrow; Magnetic Resonance Imaging
Keywords: Osteoarthritis; Knee; Bone; Bone Marrow; Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Physical Examination; Diagnostic Imaging; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Upper tibial resection pieces usually removed from patients operated for a total knee prosthesis will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee osteoarthritis: Patients with knee osteoarthritis, classified Kellgren-Lawrence 3 or 4, with asymmetric femorotibial joint space narrowing that will follow a surgery for a prosthetic replacement of the knee wil follow the following interventions:
  * Clinical evaluation
  * Radiographic assessment of osteoarthritis
  * Magnetic resonance imaging (MRI)
  * Histological evaluation of the surgical piece
  Interventions: Diagnostic Test: Clinical evaluation; Diagnostic Test: Radiology; Diagnostic Test: Dynamic contrast-enhanced magnetic resonance imaging; Diagnostic Test: Evaluation of histological status

INTERVENTIONS:
Diagnostic Test: Clinical evaluation — Functional scores for the pathological joint will be determined
Diagnostic Test: Radiology
Diagnostic Test: Dynamic contrast-enhanced magnetic resonance imaging — Patients will be examined using a 3T MR scanner (MR 750W, General Electrics, Milwaukee, WI) with a dedicated knee coil. Subchondral bone marrow vascularization in medial and lateral femorotibial compartments will be assessed with DCE-MRI and lesions will be graded on MR images.
Diagnostic Test: Evaluation of histological status — Upper tibial resection pieces will be collected and the vascularization will be determined according to the OARSI score

SUMMARY:
Patients with osteoarthritis of the knee undergo visible joint changes in radiology and Magnetic resonance imaging (MRI) tests, but also clinically and histologically. The area of greatest change is at the subchondral/cartilage bone junction.

Investigators will determine the association between preoperative clinical evaluation (IKDC and Womac scores), radiological classifications and histopathology.

In addition, the role of inflammation in the pathogenesis of osteoarthritis is being given major interest, and inflammation is closely linked with vascularization. It was recently demonstrated that dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) could identify the subchondral bone marrow vascularization changes occurring in osteoarthritis in animals.

These changes appeared before cartilage lesions were visible and were correlated with osteoarthritis severity. Thus the opportunity to obtain an objective assessment of bone vascularization in non-invasive conditions in humans might help better understanding osteoarthritis pathophysiology and finding new biomarkers. Investigators hypothesized that, as in animals, DCE-MRI has the ability to identify subchondral bone marrow vascularization changes in human osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis, classified Kellgren-Lawrence 3 or 4, with asymmetric femorotibial joint space narrowing
* Patients requiring a total knee prosthesis

Exclusion Criteria:

* Patients with a known progressive inflammatory pathology (rheumatoid arthritis,...).
* Patients with previous surgery of the knee
* Contra-indication for magnetic resonance imaging, chronic renal failure (creatinine clearance < 30 ml/min), contrast media allergy, orthopaedic hardware around the knee. Patients in whom motion artifacts impaired image analysis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis, classified Kellgren-Lawrence 3 or 4, with asymmetric femorotibial joint space narrowing, that need a knee prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Score IKDC (International Knee Documentation Committee) for functional evaluation of the articulation | At inclusion
  The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Meanwhile, the sports activity subscale focuses on functions like going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks patients one simple question: how is their knee at present versus how was their knee prior to injury?
  Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Score WOMAC (Western Ontario McMaster University ) for functional evaluation of the articulation | At inclusion
  An arthritic pain scoring system ranging from 0-no pain/disability to 100-most severe pain/disability
Radiographic assesment of osteoarthritis according to absence/presence of pathology | At inclusion
Assesment of subchondral bone marrow vascularization by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) according to the % Area Under the Curve (AUC) of perfusion value | At inclusion
The magnetic resonance imaging -based Whole-Organ Magnetic Resonance Imaging (WORMS) Score to assess the full spectrum of knee structures and the severity of knee pathologies | At inclusion
  WORMS scoring for cartilage. Cartilage lesions are scored with the WORMS system on an eight-point scale, as follows: 0 indicates normal cartilage; 1, increased signal with fluid-sensitive intermediate-weighted sequences; 2, partial-thickness defect less than 1 cm in greatest width; 2.5, full-thickness defect less than 1 cm in greatest width; 3, multiple areas of partial-thickness (grade 2) defects intermixed with areas of normal thickness or a partial-thickness defect wider than 1 cm but less than 75% of the region; 4, diffuse (≥75% of the region) partial-thickness loss; 5, multiple areas of full-thickness loss (grade 2.5) or a full-thickness defect wider than 1 cm but less than 75% of the region; and 6, diffuse (≥75% of the region) full-thickness loss.
Analysis of the surgical section by the OARSI score (Osteoarthritis research society international) for evaluation of histologic status | through study completion, an average of 3 years
  The OARSI system is based on histologic features of osteoarthritis progression. The system employs analysis of a standard block/section assessment by grade, stage of arthritis with subsequent calculation of an arthritis score. With normal cartilage as grade 0, osteoarthritis severity is divided into six grades. Grades 1-4 involve articular cartilage changes only, whereas grades 5 and 6 involve subchondral bone as well.
Osteoarthritis pathology assessment according to the number of vessels in the subchondral bone | through study completion, an average of 3 years
  Analysis of the surgical section
Osteoarthritis pathology assessment according to the thickness of the subchondral bone | through study completion, an average of 3 years
  Analysis of the surgical section

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Coursier, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille